CLINICAL TRIAL: NCT06001047
Title: Effect of Head Acupuncture on Residual Symptoms After Canalith Repositioning Procedure for Benign Paroxysmal Positional Vertigo: a Single-center Randomized Controlled Trial.
Brief Title: Head Acupuncture Treat Residual Symptoms After Canalith Repositioning Procedure for BPPV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xi'an No.3 Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACURS
Record Dates: First submitted 2023-05-11; First posted 2023-08-21 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-05

CONDITIONS: Benign Paroxysmal Positional Vertigo
MeSH Terms: conditions — Benign Paroxysmal Positional Vertigo

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (acupuncture group) (Experimental): Treatment patients with residual symptoms after successful manual repositioning by electroacupuncture
  Interventions: Procedure: Group A
- Group B (betahistine group) (Active Comparator): Treatment patients with residual symptoms after successful manual repositioning by oral betahistine
  Interventions: Drug: Group B

INTERVENTIONS:
Procedure: Group A — Acupoint selection: The location of the vertigo-auditory area follows the positioning standard of Jiao Shunfa's Head Acupuncture. Operation: Electroacupuncture stimulation in the vertigo-auditory area of affected side. Pulse electrotherapy produced by Wujin Changcheng Medical Instrument. Sparse-dense waveforms are selected, with a voltage of 2-4V, a frequency of 60-80 times/min, and the intensity is determined by the patient's tolerance. The needle is in affected side for 30 minutes, and treatment is given once daily for a total of 5 days.
  Other Names: Scalp acupuncture
  Arms: Group A (acupuncture group)
Drug: Group B — The original text is related to a medication called Pitavastatin Calcium Tablets, commonly known as "Minshilang" in Chinese, produced by Weicai (China) Pharmaceutical Co., Ltd. The dosage is 12mg, three times a day (Tid) for four consecutive weeks. Compliance monitoring is conducted by counting the remaining tablets in the medication packaging box brought by patients during the 4-week follow-up period. Concurrent use of other medications that may affect the observation results, such as anti-anxiety drugs, vestibular suppressants, and anti-dizziness Chinese patent medicines, is considered a violation of the protocol.
  Other Names: betahistine group
  Arms: Group B (betahistine group)

SUMMARY:
Benign paroxysmal positional vertigo (BPPV) is the most common peripheral vestibular disorder, and currently, manual repositioning techniques are often used for treatment. However, up to 30%-50% of patients may experience residual symptoms such as non-rotational dizziness, heaviness, instability, and emotional disturbances even after successful repositioning, which significantly impacts their daily functioning and quality of life. Electroacupuncture therapy has been proven to be an effective treatment for dizziness and has been applied to various vestibular disorder patients. However, the efficacy of electroacupuncture on the residual effects of successfully repositioned BPPV patients remains unclear. This study aims to explore the effectiveness of three regimens: electroacupuncture, betahistine in patients with residual symptoms after successful manual repositioning.

DETAILED DESCRIPTION:
Research objectives:

1. Explore the risk factors that influence residual effects after BPPV and develop a predictive score chart.
2. Determine the gait characteristics of patients with residual effects after successful repositioning of BPPV.
3. Compare the clinical efficacy of different intervention strategies for the treatment of residual symptoms after successful repositioning of BPPV.

Research subjects:

From June 2023 to June 2024, patients aged between 18-65 who are first diagnosed with BPPV will be recruited from the outpatient and inpatient departments of the Third Hospital of Xi'an City, affiliated to Northwest University. For posterior canal BPPV, Epley or Semont maneuver will be performed; for horizontal canal BPPV, Gufoni maneuver will be performed; for anterior canal BPPV, Yacovino maneuver will be performed. The patients will be observed for 30 minutes after the positioning maneuver to confirm the successful repositioning. On the second day after the maneuver, the follow-up personnel of the research team will contact the patient by phone or online to determine whether they have residual dizziness symptoms and whether they are willing to participate in the study. Those who agree can come to the hospital for reassessment to confirm the successful repositioning.

Residual symptom evaluation criteria:

On the 2nd day after successful repositioning, ask the patient if they have persistent nonspecific symptoms such as dizziness, feeling of heaviness in the head, unsteadiness, or floating sensation, without positional vertigo.

Sample size estimation:

According to the sample size design plan of randomized controlled studies, with a Type I error of α=0.05, a Type II error of 1-β=0.8, an incidence rate of P1=0.6 in the intervention group, an incidence rate of P2=0.45 in the control group, and a 1:1 ratio, 50 participants are allocated to each group with a total of 150 participants. Assuming a certain proportion of dropouts in each group, the sample size of each group required for enrollment is 60 participants.

Randomization and blinding:

The postoperative patients were randomly divided into two groups: Group A (acupuncture group) and Group B (betahistine group) using SPSS 20.0 software. This study did not apply blinding to the operators or patients, while the outcome assessors and data analysts were blinded.

Data collection: Baseline data including demographic information, medical history, physical examination, laboratory tests, and vestibular function tests were collected at enrollment. Dizziness Handicap Inventory (DHI) and Visual Analog Scale (VAS) scores were collected at baseline, 3 days after treatment, 1 week after treatment, 2 weeks after treatment, and 4 weeks after treatment. In addition, balance function and gait tests were performed at each time point.

ELIGIBILITY:
Inclusion Criteria:

1. According to the diagnostic criteria and therapeutic efficacy evaluation for benign paroxysmal positional vertigo (BPPV) formulated by the Otolaryngology-Head and Neck Surgery Branch of the Chinese Medical Association, the patient was confirmed as having BPPV and the repositioning maneuver was successful.
2. After the maneuver, the patient's clinical symptoms were relieved, with no sense of rotation or dizziness, but residual symptoms such as discomfort and unsteady gait persisted.
3. There were no obvious communication barriers or visual impairments.
4. The patient and their family members agreed to the treatment plan.

Exclusion Criteria:

* Patients with other ear diseases, history of head trauma or surgery;

  * Patients who are weak and unable to tolerate, pregnant women;

    * Patients who have undergone vestibular rehabilitation training before this treatment; ④ Patients with joint diseases that affect balance and walking; ⑤ Patients with a history of brain organic diseases (such as tumors, stroke, cerebral hemorrhage) or severe neurological diseases; ⑥ Patients with incomplete data or who withdraw from treatment midway.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) score | 1weeks after treatment
  A scale used to evaluate the degree of dizziness in patients, scores range from 0 to 10, with higher scores indicating more severe degree of dizziness they feel.
Dizziness Handicap Inventory | 1weeks after treatment
  Self-perceived handicapping effects imposed by dizziness. Internal consistency (Cronbach's alpha: 0.92), Test-retest reliability r = 0.95

SECONDARY OUTCOMES:
Foam posturography | 1weeks after treatment
  The sponge-cushion posturing is a quantitative method for measuring postural stability. The test-retest reliability of sponge-cushion posturing is good (ICC = 0.887-0.973)

CONTACTS AND LOCATIONS:
Overall Officials: Mingze Zhao, PhD, Study Chair — Xi'an No.3 Hospital
Locations (1):
- Xi'an No3 Hospital, Xi'an, China

IPD SHARING:
Plan to Share IPD: No